CLINICAL TRIAL: NCT01562288
Title: Adjuvant Chemotherapy Combined With Trastuzumab in the Randomized Phase III Trial N9831 Actively Immunizes Patients Against Tumor Antigens
Brief Title: Studying Blood and DNA Samples From Patients With Breast Cancer Treated With Chemotherapy With or Without Trastuzumab
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-N9831D-NCCTG-ICSC; NCI-2012-00687 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000726841 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; HER2-negative breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum and DNA extracted from peripheral blood mononuclear cell samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Previously collected serum and DNA from peripheral blood mononuclear cell samples are analyzed for HER2-specific antibodies and FcγR genotype by ELISA and PCR.
  Interventions: Genetic: DNA analysis; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Other: enzyme-linked immunosorbent assay
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and DNA in the laboratory from patients who received chemotherapy with or without trastuzumab may help doctors learn more about the effects of trastuzumab on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research trial studies blood and DNA samples from patients with breast cancer treated with chemotherapy with or without trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the role of trastuzumab in the generation of HER2-specific antibodies in breast cancer patients undergoing adjuvant combination therapy.
* To determine whether the improved disease-free period and overall survival of patients treated in the adjuvant setting with combination of chemotherapy and trastuzumab is dependent on the Fcγ receptor genotype of the patient.

OUTLINE: Previously collected serum and DNA samples are analyzed for HER2-specific antibodies and FcγR genotype by enzyme-linked immunosorbent assay (ELISA) and polymerase chain reaction (PCR).

ELIGIBILITY:
• Patients with HER-2-overexpressing node-positive or high-risk node-negative breast cancer enrolled on NCCTG-N9831

* Pre- and post-treatment serum and DNA samples of patients treated with doxorubicin and cyclophosphamide followed by paclitaxel with or without trastuzumab (Herceptin®)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on NCCTG-N9831.
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
disease-free survival | up to 1 month
overall survival | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Keith L. Knutson, MD, PhD, Principal Investigator — Mayo Clinic